CLINICAL TRIAL: NCT05413629
Title: The Effect of Web Based Education on the Treatment Process of Women Undergoing Intrauterine Insemination (IUI) on the Level of Coping With Infertility Stress and Infertility Self-Efficacy
Brief Title: The Effect of Web Based Education on the Level of Coping With Infertility Stress and Infertility Self-Efficacy
Acronym: education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Duzce U; hilalkaradeniz1 (Other: Health Science Faculty)
Record Dates: First submitted 2022-05-09; First posted 2022-06-10 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Infertility, Female; Educational Problems; Intrauterine Insemination
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: Solomon four-group, randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group1 (n=33) (No Intervention): Control 1: Pretest negative and post test positive group
- Group 2 (n=33) (No Intervention): Control 2: Pretest positive and post test positive
- Group 3 (n=33) (Experimental): Experimental 1: Pretest negative and post test positive
  Interventions: Other: Web-based patient education for the intrauterine insemination (IUI) treatment process
- Group 4 ( n=33) (Experimental): Experimental 2: Pretest positive and post test positive
  Interventions: Other: Web-based patient education for the intrauterine insemination (IUI) treatment process

INTERVENTIONS:
Other: Web-based patient education for the intrauterine insemination (IUI) treatment process — Web-based training is 60 minutes in total, including 4 modules. The web-based training content includes general information about fertility, infertility diagnosis-treatment methods, drugs used in IUI treatment and its application, and issues to be considered after IUI.
  Arms: Group 3 (n=33); Group 4 ( n=33)

SUMMARY:
In the study, it is aimed to reduce the infertility stress level of women undergoing infertility treatment, to increase the level of coping with infertility stress, to increase infertility self-efficacy, to evaluate the usability of web-based education in the field of infertility, to increase the effectiveness and quality of education by integrating web-based education into the nursing care process, and continuous traceability, to prevention of possible wrong treatment process management in the field of infertility, to prevention of possible loss of cycles and to prevention the material and moral couple from being adversely affected by this process.

Method: The study was planned to be carried out between 20.01.2022 and 01.06.2023 with women between the ages of 23-39 who applied to Düzce University Health Practice and Research Center, Infertility Polyclinic. In the research, the Solomon four-group design sample design consisting of two experimental and two control groups will be used. The study planned to consist of a total of 132 patients, 33 patients in each group, taking into account possible data losses. By design, all of the pre-test and post-test measurement tools will be applied to the first experimental and control group, and only the post-test measurement tools will be applied to the second experimental and control group. Randomization will be applied in determining the experimental and control groups. The data will be collected using Personal Information Form (Appendix-1), Infertility Stress Scale (ISS) (Appendix 2), Coping with the Infertility Stress Scale (CISS) (Appendix-3), and Infertility Self-Efficacy Scale - Short Form (ISE-SF) (Appendix 4). Research data will be collected in approximately day 24 to 27 days for each patient from the initiation of Controlled Ovarian Stimulation (COS) treatment to pregnancy determination of patients planned for intrauterine insemination (IUI) treatment.

Web-based training is 60 minutes in total, including 4 modules. The web-based training content includes general information about fertility, infertility diagnosis-treatment methods, drugs used in IUI treatment and its application, and issues to be considered after IUI.

DETAILED DESCRIPTION:
Infertility is defined as the inability to conceive or to continue the pregnancy, despite having unprotected sexual intercourse at least twice a week for a year and at least twice a week. It is reported that more than 80 million people around the world are unable to have children due to medical reasons, and 15% of couples in Turkey are diagnosed with infertility. When we look at the literature, it is suggested that infertility and assisted reproduction treatments cause an increase in the level of stress, depression and anxiety in individuals and that it is necessary to strengthen their coping with this process.

Aim: This study was planned as a randomized controlled experimental study in order to examine the effect of web-based education about the treatment process on the level of coping with infertility stress and infertility self-efficacy to women undergoing Intrauterine Insemination (IUI) treatment.

Objective: In the study, it is aimed to reduce the infertility stress level of women undergoing infertility treatment, to increase the level of coping with infertility stress, to increase infertility self-efficacy, to evaluate the usability of web-based education in the field of infertility, to increase the effectiveness and quality of education by integrating web-based education into the nursing care process, and continuous traceability, to prevention of possible wrong treatment process management in the field of infertility, to prevention of possible loss of cycles and to prevention the material and moral couple from being adversely affected by this process.

Method: The study was planned to be carried out between 20.01.2022 and 01.06.2023 with women between the ages of 23-39 who applied to Düzce University Health Practice and Research Center, Infertility Polyclinic. In the research, the Solomon four-group design sample design consisting of two experimental and two control groups will be used. Power analysis (G*Power 3.1.9.2) was performed on the basis of a previous similar research in the selection of the sample. Accordingly, the sample of the study was planned to consist of a total of 132 patients, 33 patients in each group, taking into account possible data losses. By design, all of the pre-test and post-test measurement tools will be applied to the first experimental and control group, and only the post-test measurement tools will be applied to the second experimental and control group. Randomization will be applied in determining the experimental and control groups. The data will be collected using Personal Information Form (Appendix-1), Infertility Stress Scale (ISS) (Appendix 2), Coping with the Infertility Stress Scale (CISS) (Appendix-3), and Infertility Self-Efficacy Scale - Short Form (ISE-SF) (Appendix 4). The preliminary application of the research will be completed with an average of 16 women, who constitute at least 10% of the sample of 132 people. Research data will be collected in approximately day 24 to 27 days for each patient from the initiation of Controlled Ovarian Stimulation (COS) treatment to pregnancy determination of patients planned for intrauterine insemination (IUI) treatment.

In the research, the experimental group will be given a brief face-to-face briefing about the treatment process as well as a detailed training via the website. Web-based training is 60 minutes in total, including 4 modules. The web-based training content includes general information about fertility, infertility diagnosis-treatment methods, drugs used in IUI treatment and its application, and issues to be considered after IUI. The patients in the control group, on the other hand, will be given the hospital's drug administration brochure after brief face-to-face information and no other intervention will be made. When the patients come back to the hospital for IUI treatment, they will fill out the Infertility Stress Scale (ISS), Coping with the Infertility Stress Scale (CISS), Infertility Self-Efficacy Scale - Short Form (ISE-SF). BHCG results of the patients will be learned on the 14th day after IUI.

ELIGIBILITY:
Inclusion Criteria:

* Applying to Düzce University Health Practice and Research Center Infertility Polyclinic
* Primary infertility,
* Controlled Ovarian Hyperstimulation (COH) planned for the treatment of intrauterine insemination (IUI),
* Having the equipment (mobile phone, computer, tablet, internet) to access web-based education,
* No chronic disease,
* No diagnosed psychiatric disease,
* Agreeing to participate in the research,
* Having the ability to understand and comprehend the questionnaires

Exclusion Criteria:

* Controlled Ovarian Hyperstimulation (COH) is not planned in the treatment of intrauterine insemination (IUI),
* Give up treatment,
* Not having the equipment (mobile phone, computer, tablet, internet) to access web-based education,
* Having a chronic disease,
* Having a diagnosed psychiatric disease,
* Those who do not agree to participate in the research,
* Those who do not have the ability to understand and comprehend the questionnaires

Ages: 23 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Infertility Stress Scale | 24 to 27 days
  The level of infertility stress assessed by Infertility Stress Scale (ISS). The scale consists of 3 sub-dimensions. The total minimum score that can be obtained from the scale is 0 and the total maximum score is 46. As the score obtained from the scale increases, the stress level of the individual increases and as the score decreases, the stress level decreases.
Coping with the Infertility Stress Scale | 24 to 27 days
  The level of coping with infertility stress assessed by Coping with the Infertility Stress Scale (CISS). The scale consists of 4 sub-dimensions. The total minimum score that can be obtained from the scale is 19 and the total maximum score is 74. As the score obtained from the scale increases, the individual copes better with stress, and as it decreases, the individual copes less well.

SECONDARY OUTCOMES:
Infertility Self-Efficacy Scale - Short Form | 24 to 27 days
  The level of infertility self-efficacy assessed by ISE-SF (Infertility Self-Efficacy Scale - Short Form). The minimum score that can be obtained from the scale is 8 and the maximum score is 32. Higher scores indicate higher self-efficacy and lower scores indicate lower self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Nurdan Demirci, Prof., Study Director — Duzce University
Locations (1):
- Hilal Karadeniz, Düzce, Turkey (Türkiye)

REFERENCES:
- [Derived] Yalazi RO, Demirci N. The effect of bladder training with mobile application on quality of life and sexual satisfaction in women with overactive bladder: randomized controlled study. World J Urol. 2025 Sep 25;43(1):573. doi: 10.1007/s00345-025-05917-6. PMID 40996496